CLINICAL TRIAL: NCT06397391
Title: Nonlinear Absorber in Essential Tremor Treatment
Acronym: TREM-AB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL21_0984
Record Dates: First submitted 2022-05-23; First posted 2024-05-02 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Essential Tremor
Keywords: Essential tremor; Passive treatment; Nonlinear absorber
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical device (Experimental): Patients will test medical device on site during 1 hour. EMG (electromyogram) and accelerometry will be performed before and after this hour. As same as clinical scale (Fahn-tolosa-Marin)
  Interventions: Device: TREM-AB

INTERVENTIONS:
Device: TREM-AB — Wearing medical device on site during 1 hour

SUMMARY:
The goal of this study is to develop a non linear absorber for patients with essential tremor (ET). It 's an extern passive medical device which should improve patients tremor.

Investigators will evaluate the impact of this medical device through one clinical scale (Fahn-Tolosa-Marin) and accelerometry record. Investigators focus on motor improvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult man or woman between 20 and 90 years old
* Diagnosis of ET (Essential Tremor) established by a neurologist
* ET affecting the upper limbs, associated or not with head tremor
* Drug-resistant nature of ET (failure of beta-blockers, mysoline, benzodiazepine)
* Affiliate to a social security or similar system
* Having given written consent to participate in the study, free and informed.

Exclusion Criteria:

* Severe comorbidity
* ET affecting only the leader
* Wounds on the forearm
* Modification of treatment or surgery to manage ET, planned within 3 months following inclusion
* Cognitive disorder known or suspected by the investigator
* Pregnant or breastfeeding woman
* Persons placed under guardianship, curatorship or under judicial protection
* Persons deprived of liberty, subject to psychiatric care or admitted to a health or social establishment for purposes other than that of clinical investigation

Criteria for premature discharge

* MMSE (Mini-Mental State Examination) score<24;
* ET of the patient with frequency range not between 4 to 6 Hz or 8 to 12 Hz and/or amplitudes of movement greater than 20°.
* modification of treatment for ET or performance of tremor surgery before the final visit;
* withdrawal of consent or refusal to continue visits.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Tremor improvement | 6 months maximum
  To assess tremor improvement, investigators will use the Fahn-Tolosa-Marin rating scale. This scale allows, thanks to a score, to assess clinical and functional evaluation of the tremor. Different aspect of the tremor are evaluate like the frequency of the tremor of the head, hand, arm..etc. and the impact of the tremor on daily actions (like writing, drawing, …).
  This score will be assessed at Visit 1 and 2. During visit 2, the assessment will be performed before and 1 hour after wearing the device.

SECONDARY OUTCOMES:
Tremor frequency | 6 months maximum
  To assess tremor frequency, investigators will use accelerometry record and electromyography.
  This score will be assessed at Visit 1 and 2. During visit 2, the assessment will be performed before and 1 hour after wearing.the device.
Tolerance to wearing the device | 6 months maximum
  Adverse reactions occurring during use of the device
Patient satisfaction with the device measured by a specific multidimensional questionnaire | 6 months maximum
  A multidimensional questionnaire has been built specifically for the study. An EVA scale is used to assess whether the patient has experienced discomfort, pain or discomfort (0-10). The higher the score, the more severe the discomfort.
  Ease of installation of the device and intention to use it on a daily basis if this was possible are evaluated by questions with binary responses (yes or no).
  Free fields are used to complete these responses and to suggest improvements of the prototype.
  This score will be assessed at the end of Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane THOBOIS, MS, PhD, Principal Investigator — Hopital neurologique Pierre Wertheimer
Locations (1):
- Service Pathologies du mouvement et neuromusculaire, Hopital neurologique Pierre Wertheimer, Bron, France

IPD SHARING:
Plan to Share IPD: No